CLINICAL TRIAL: NCT07199816
Title: The Analgesic Effect of Caudal Epidural Versus Combined Lumbar Sympathetic Block With Caudal Epidural in Patients Undergoing Redo Lumbar Surgery: A Randomized Double Blinded Controlled Trial.
Brief Title: Pain Control With Caudal Epidural vs. Combined Caudal Epidural and Lumbar Sympathetic Block .
Acronym: CLEARS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebatullah Mohammed Abdelmageed (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Hebatullah Mohammed Abdelmageed, Hebatullah Mohammed Abdelmageed, Principle Investigator, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N- 26- 2024/ MD
Record Dates: First submitted 2025-09-14; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-03

CONDITIONS: Pain Management After Surgery
Keywords: pain control
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Active Comparator): Group C (n=32): this group will receive fluoroscopy guided caudal epidural block.
  Under fluoroscopic guidance and the patients in prone position, caudal epidural injection will be achieved. A pillow will be inserted under the pelvic bones for better exposure and accessibility of thesacral hiatus. Betadine will be used for sterilization of the sacrococcygeal area and palpation of the coccygeal tip. Upon localization of the sacral hiatus, a 22-gauge, 3.5-inch length spinal needle (Spinocan®, BRAUN, Melsungen, Germany) with the image intensifier will be used to inject 1 mL of contrast media (Omnipaque 300; GE Healthcare, Carrigtohill, Co. Cork, Ireland). After confirming the right needle position and excluding intravascular, intrathecal, and soft tissue infiltration, 10 cc of the treatment drug (8 ml of 0.5%lidocaine mixed with 2ml of 8 mg dexamethasone) will be injected.
  Interventions: Procedure: Fluoroscopy-Guided Caudal Epidural Block
- Group LC (Active Comparator): Group LC: Group (n=32): this group will receive combined fluoroscopy guided caudal epidural block and lumbar sympathetic ganglion block.
  Under fluoroscopic guidance, LSGB will be performed. The block level and side will be determined. Patients will be kept in the prone position while C-arm (GE OEC 9900 C- of the anteroposterior, oblique, and lateral view are examined to verify the correct entrance sit. The skin will be prepared in an aseptic manner. Approach the anterolateral border of the inferior sec of the L2 vertebral body or the upper portion of the L3 vertebral body of the affected side where the pain exists, using a 21-gauge Chiba needle.
  Following the confirmation of the needle location via fluoroscopic imaging, an aspiration test will be performed in order to rule out the presence of blood, following by injection of a contrast medium. Following that, 2 mL of 8mg dexamethasone will be diluted with 8 mL of 1% lidocaine and injected unilaterally at one level.
  Interventions: Procedure: Combined Lumbar Sympathetic Ganglion Block and Caudal Epidural Block

INTERVENTIONS:
Procedure: Fluoroscopy-Guided Caudal Epidural Block — Under fluoroscopic guidance, the patient in the prone position will receive a caudal epidural injection through the sacral hiatus. A 22-gauge, 3.5-inch spinal needle (Spinocan®, BRAUN) is used to inject 1 mL of contrast media (Omnipaque 300) to confirm correct needle placement. Then, 10 mL of treatment solution (8 mL of 0.5% lidocaine and 2 mL of 8 mg dexamethasone) is administered.
  Arms: Group C
Procedure: Combined Lumbar Sympathetic Ganglion Block and Caudal Epidural Block — Patients will receive both a caudal epidural block and a lumbar sympathetic ganglion block (LSGB) under fluoroscopic guidance. The LSGB is performed at the L2 or L3 vertebral body on the affected side using a 21-gauge Chiba needle. After confirming needle position with contrast imaging, 10 mL of solution (2 mL of 8 mg dexamethasone + 8 mL of 1% lidocaine) is injected. A caudal block is then performed as described above.
  Arms: Group LC

SUMMARY:
Comparing the analgesic effect of caudal epidural versus combined lumbar sympathetic block with caudal epidural in patients undergoing redo spinal surgery.

DETAILED DESCRIPTION:
To evaluate the improvement in pain score using numerical rate scale (NRS) over 4 months and compare this between the two groups.

* To assess and compare the improvement of motor activity and early ambulation using EuroQo lmeasure (EQ-5D) between the two groups.
* To evaluate and compare the overall patient satisfaction between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I to III.
* Undergoing lumbar spine surgery level L4-5/ L5-S1 for the second time.
* Duration of chronic low back pain > 3months.

Exclusion Criteria:

* Emergency surgeries.
* Bleeding disorder.
* patient refusal for the procedure.
* Pregnancy.
* Neoplastic diseases, allergies to contrast.
* Liver failure or kidney failure .

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (Numerical Rating Scale - NRS) | over 3 months postoperative
  Pain intensity will be assessed using the Numerical Rating Scale (NRS), where patients rate their pain from 0 (no pain) to 10 (worst possible pain). NRS scores will be compared between the two groups (caudal epidural block vs. combined lumbar sympathetic and caudal epidural block) to evaluate the long-term effectiveness of the interventions.

SECONDARY OUTCOMES:
Postoperative pain intensity (NRS) | over 24 hours after surgery
  Pain will be measured using the Numerical Rating Scale (NRS), where 0 = no pain and 10 = worst pain imaginable. Pain scores will be recorded preoperative and at 6, 12, 18, and 24 hours postoperatively to assess short-term pain control.
Time to first postoperative analgesic request | postoperative period up to hospital discharge
  Time (in hours) from the end of the procedure to the first request for analgesia. A longer time indicates more effective initial pain relief.
Total postoperative morphine consumption | postoperative period up to hospital discharge
  Total amount of morphine administered postoperatively will be recorded in milligrams to evaluate analgesic requirement across both groups.
Long-term pain relief using WHO pain relief criteria | over 3 months after the procedure
  Pain relief will be categorized based on WHO four-grade scale: Complete Remission (CR), Partial Remission (PR), Mild Remission (MR), and No Response (NR), assessed at 3 months to evaluate long-term analgesic effect.
Functional recovery and ambulation (EuroQol) | over 3 months postoperative
  The EuroQol (EQ-5D) questionnaire will be used to assess functional status and early ambulation at multiple follow-up points. Higher scores reflect better recovery and quality of life.
Length of hospital stay | From admission to discharge
  Total number of days the patient remains hospitalized will be recorded to evaluate the effect of the intervention on recovery time.
Incidence of complications related to the blocks | Intraoperative and postoperative period up to hospital discharge
  Any adverse events or complications related to caudal epidural or lumbar sympathetic ganglion blocks (e.g., infection, hematoma, neurologic symptoms) will be recorded and compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al-Ainy Medical School, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Participant privacy and confidentiality concerns; data sharing is not permitted under institutional policy.

REFERENCES:
- See also: Related Info — https://medicine.cu.edu.eg/